CLINICAL TRIAL: NCT00456313
Title: Rationale for Therapy With Low Dose Steroids Combined With Long-acting beta2-agonists in Patients With Allergic Asthma: Redirecting Innate Immune Responses by Long-term Treatment With High Doses of Inhaled Steroids
Brief Title: No Resistance After Long Term Treatment SERETIDE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of data
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM109352
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: asthma; fluticasone propionate; salmeterol/fluticasone propionate; combination product; innate immune response; neutrophil priming
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- arm 1 (Active Comparator)
  Interventions: Drug: FLIXOTIDE and SERETIDE

INTERVENTIONS:
Drug: FLIXOTIDE and SERETIDE — comparator

SUMMARY:
This multi centre, double blind, comparator controlled, parallel group study is to determine whether asthma treatment with high doses of fluticasone propionate (FP) redirects a Th2/ eosinophil response towards a more treatment resistant neutrophil/ monocyte response and whether this occurs to a lesser extent in asthmatic subjects treated with the combination product of salmeterol and fluticasone propionate (SFC). The primary endpoint is the mean change in priming of blood neutrophils assessed by marker A17. After a run-in period of 4 weeks subjects will enter a 24 weeks high dose treatment (FP 500 mcg bd) or a 12 week medium-dose treatment with FP 250 mcg bd followed by a 12 week treatment with SFC 50/ 250 mcg. At the visits lung function measurements, ACT, eNO measurements and a blood sample will be performed. A total of 50 randomised subjects are planned to be recruited in this study

ELIGIBILITY:
Inclusion:

* Positive skin prick test
* History of asthma (GINA)
* Regular treatment with FP with/without LABA at least 4 weeks before visit 1
* History of recurrent episodes of wheezing, breathlessness, chest tightness and/ or coughing in the previous year.
* Able to use a DISKUS™ inhaler
* Able perform reproducible lung function tests at Visit 1

Inclusion criteria treatment period:

* FEV1 % predicted > 70%
* ACT score < 25 after run-in period

Exclusion criteria run-in period:

* Hospitalised for asthma within 4 weeks prior to Visit 1
* Acute upper respiratory tract infection or a lower respiratory tract infection within 4 weeks prior to Visit 1
* Oral, parental or depot corticosteroids within 4 weeks prior to Visit 1
* Hepatic impairment or other significant disease

Exclusion criteria treatment period:

* Non-compliance (< 70%)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Estimated); Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in neutrophil priming in blood as assessed by marker A17 | on going

SECONDARY OUTCOMES:
Activation in markers such as A27, CD11b, L-selection, CD16, CD32, VLA-4 and CD66b in whole blood- Cytokine/chemokine determination by multiplex assay in cell free serum- Asthma control measured - Lung function: FEV1, FVC and PEF- eNO | on going

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Utrecht, Netherlands